CLINICAL TRIAL: NCT04837287
Title: Investigation of the Effect of Short and Long Term Stretching Exercise on Muscle Elasticity in Two Different Muscle Groups
Brief Title: Investigation of the Effect of Different Term Stretching Exercise on Muscle Elasticity in Two Different Muscle Groups
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Eda Tonga, Assoc. Prof., Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2020.47
Record Dates: First submitted 2021-02-21; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Rehabilitation; Muscle Tightness
Keywords: Static Stretching Exercises; Stretching Time; Muscle Elasticity; Muscle Flexibility

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants of the study will be included in the stretching exercise program, but the participants will not have information about which group the participants belong to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Stretching Exercise for 10 Seconds (Active Comparator): After the participants are given one session of training, the participants do the exercises themselves at home.
  Interventions: Other: Static Stretching Exercise for 10 Seconds
- Static Stretching Exercise for 30 Seconds (Active Comparator): After the participants are given one session of training, the participants do the exercises themselves at home.
  Interventions: Other: Static Stretching Exercise for 30 Seconds

INTERVENTIONS:
Other: Static Stretching Exercise for 10 Seconds — The participants were asked to do a static stretching exercise for the Hamstring and Gracilis muscles for 10 seconds. The participants were asked to continue for 8 weeks, 3 days a week, 3 times a day - 10 repetitions.
  Arms: Static Stretching Exercise for 10 Seconds
Other: Static Stretching Exercise for 30 Seconds — The participants were asked to do a static stretching exercise for the Hamstring and Gracilis muscles for 30 seconds. The participants were asked to continue for 8 weeks, 3 days a week, 3 times a day - 10 repetitions.
  Arms: Static Stretching Exercise for 30 Seconds

SUMMARY:
In the literature, the evidence regarding the effects of different static stretching times on elasticity is very limited, and the evidence on the effects on flexibility varies. Although 10 to 30 seconds of static stretching is said to be effective, studies on which duration is effective for which muscle group are quite limited. Based on these, the aim of this study is to examine the effects of stretching exercises of different periods on muscle elasticity to be applied to thin and thick muscle groups. In order to evaluate its effectiveness, assessment of evaluation of muscle flexibility, active-passive range of motion were being applied.

DETAILED DESCRIPTION:
Flexibility, the most important component of physical fitness, is defined as the maximal range of motion occurring in the joint or joint group. Elasticity is the ability of the structure to change its shape and size with the effect of force and to return to its previous position when the force is removed. These two components are also very effective on strength, agility, balance, speed, coordination and proprioception, which are other components of physical fitness. It is very important in reducing stress and tension, relieving muscle cramps, muscle relaxation, body fitness, reducing risks of injury and pain, regular sleep and daily life activities. Good levels of this increase the efficiency of the movement.

Different stretching protocols are applied in traditional rehabilitation to increase these levels. Static stretching, which is one of these stretching protocols, is known to prevent injuries and benefit performance as a result of increasing the range of motion. It is a type of stretching that minimizes the risk of injury as well as easy application. However, stretching times that will change the elasticity and flexibility of a large-thick muscle and a thin-long muscle are different. In the literature, the evidence regarding the effects of different static stretching times on elasticity is very limited, and the evidence on the effects on flexibility varies. Although 10 to 30 seconds of static stretching is said to be effective, studies on which duration is effective for which muscle group are quite limited.

Based on these, the aim of our study is to examine the effects of stretching exercises of different periods on muscle elasticity to be applied to thin and thick muscle groups. The study will be carried out on healthy, sedentary people aged 20-45 years. People who agree to participate in the study will be randomly divided into two groups. Static stretching will be applied to the hamstring and gracilis muscles of one group for 10 seconds while static stretching will be applied to the other group for 30 seconds. Static stretching exercises will be applied 8 weeks, 3 days a week, 3 times a day in 10 repetitions. On the dominant legs of the participants will be evaluated muscle elasticities with Myoton, muscle flexibility with flexibility tests, joint range of motion with goniometer. As a result of our thesis study, the investigators aim to find out how many seconds of static stretching will be more effective in different muscle groups, how different stretching times will change the muscle elasticity in different muscle groups, and thanks to this information, the investigators will be more successful in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-45
* Have not had any disability or surgery in the past 6 months
* Not exercising regularly in the last 6 months
* No neural signs
* To participate regularly in the study

Exclusion Criteria:

* Exercising regularly in the last 6 months,
* Having any disability or surgery not allowing stretching exercise,
* Having hip-knee-waist problem
* Having comorbidities not allowing stretching exercise such as inflammatory rheumatic disease, orthopedic and neurological disease

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Elasticity of the Muscle | Pre exercise and Week 8
  The method of measurement consists of recording damped natural oscillation of soft biological tissue in the form of an acceleration signal and the subsequent simultaneous computation of the parameters of State of Tension, Biomechanical and Viscoelastic properties. Damped natural oscillation is induced by an exterior, low force quick-release mechanical impulse under constant pre-load. At the end of this measurement, information about the muscle elasticity in logarithmic decrement on muscle is obtained. In our study, this measurement will be evaluated with Myoton.

SECONDARY OUTCOMES:
Tone of the Muscle | Pre exercise and Week 8
  The method of measurement consists of recording damped natural oscillation of soft biological tissue in the form of an acceleration signal and the subsequent simultaneous computation of the parameters of State of Tension, Biomechanical and Viscoelastic properties. Damped natural oscillation is induced by an exterior, low force quick-release mechanical impulse under constant pre-load. At the end of this measurement, information about the muscle tone in Hz is obtained. In our study, this measurement will be evaluated with Myoton.
Stiffness of the Muscle | Pre exercise and Week 8
  The method of measurement consists of recording damped natural oscillation of soft biological tissue in the form of an acceleration signal and the subsequent simultaneous computation of the parameters of State of Tension, Biomechanical and Viscoelastic properties. Damped natural oscillation is induced by an exterior, low force quick-release mechanical impulse under constant pre-load. At the end of this measurement, information about the muscle stiffness in N/m is obtained. In our study, this measurement will be evaluated with Myoton.
Demographic Data Form | Pre exercise
  The participants are asked to fill in an information form that evaluates age, gender, educational background, occupation, presence of permanent disease, disability or surgeries, and when it happened, whether there are hip-knee-waist problems.
Hamstring Muscle Flexibility | Pre exercise, Measurement for 7 weeks, Week 8
  The Hamstring muscle is evaluated by the Sit - Lie test. The participants are asked to take off their shoes and sit on the floor and place the soles flat on the measuring board. The participants are asked to lie forward as far as the participants can reach their fingertips by moving their bodies forward without bending the participants's knees and waiting at least 2 seconds at the last point. The point where the participants can reach is marked and the distance between the level of the feet and the marked point is measured by tape measure. The measurement is repeated twice and the highest value is recorded in cm.
Gracilis Muscle Flexibility | Pre exercise, Measurement for 7 weeks, Week 8
  The Gracilis muscle is evaluated by Hip Abduction Flexibility Test. For testing, the participants sits with hip abduction, flexion and external rotation, knees flexed, and feet soles adjacent. The participants is asked to push their knees down, holding their knees. The distance between the lateral condyle of both knees and the ground is measured by tape measure. The measurement is recorded in cm.
Active - Passive Joint Range of Motion | Pre exercise, Measurement for 7 weeks, Week 8
  The measured joint is placed according to the anatomical position, and this position is considered the starting position, and the measurement starts here. The participants is asked to do the movement as much as the participants can, and an angle measurement is made. In our study, this measurement will be done with the universal goniometer.
Exercise Diary | Pre exercise, Measurement for 7 weeks, Week 8
  The participants will note the number of exercises the participants did at home in the exercise diary next to the image showing the exercise example day by day. All exercises will be evaluated as 100% when done with the number of repetitions required.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Dilge AŞIK, PT, Principal Investigator — Marmara University Faculty of Health Sciences; Eda TONGA, Assoc. Prof., Study Director — Marmara University Faculty of Health Sciences; Yavuz YAKUT, Prof. Dr., Study Director — Hasan Kalyoncu University Faculty of Health Sciences
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)